CLINICAL TRIAL: NCT05205798
Title: The Effect of Plate Size on Food Consumption Amount and Satiety in Healthy Women
Brief Title: The Effect of Plate Size on Food Consumption and Satiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Seliz Bağcılar, Principal Investigator, Eastern Mediterranean University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: EMU-ETK00-2020-0242
Record Dates: First submitted 2021-12-19; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Satiety; Food Consumption

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Food consumption using plates with a diameter of 23 cm first then using plates with a diameter of 31 cm
  Interventions: Behavioral: Food consumption using plates with a diameter of 23 cm.; Behavioral: Washout period; Behavioral: Food consumption using plates with a diameter of 31 cm.

INTERVENTIONS:
Behavioral: Food consumption using plates with a diameter of 23 cm. — In the experiment, individuals will consume the amount of pasta with sauce offered in the open buffet in the amount they will determine (ad libitum), using plates with a diameter of 23 cm.
Behavioral: Washout period — No interventional food consumption for 1 week
Behavioral: Food consumption using plates with a diameter of 31 cm. — In the experiment, individuals will consume the amount of pasta with sauce offered in the open buffet in the amount they will determine (ad libitum), using plates with a diameter of 31 cm.

SUMMARY:
In this study, it was aimed to investigate the effect of plate size on food consumption and satisfaction levels in healthy women.

DETAILED DESCRIPTION:
The effect of plate size on food consumption and satisfaction levels in healthy women aged between 19-35 years will be evaluated in this study. In addition to this, the relationship between the amount of food that women eat and their feelings of satisfaction will be evaluated. During the experiment, the individuals will be asked to consume the pasta with sauce which is offered in the open buffet in the amount of their own determination (ad libitum) using different sized (23 cm and 31 cm) plates. The size of the plates that individuals will use on different experimental days was determined randomly.

ELIGIBILITY:
Inclusion Criteria:

* having a score of <20 from EAT-26 test,
* not smoking,
* not following any diet,
* not having a diagnosis of any metabolic disease,
* not being color blind,
* not being a professional athlete,
* not using nutritional supplements,
* not having any food allergy,
* not being selective towards certain food.
* not being pregnant or lactating,
* not using any medication that affects appetite and body weight,
* not having the habit of consuming regular main meals.

Exclusion criteria: Failing to meet the inclusion criteria

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-01-30 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Ad libitum food intake | 30 minutes
  Measuring consumed food
Self reported mood score by Visual Analogue Scale | Baseline
  Measuring mood (from 0mm - 100mm)
  Choosing 0mm means less feeling of the emotion asked while choosing 100mm means more feeling of the emotion asked.
Self reported hunger and satiety score by Visual Analogue Scale | Baseline to 180 minutes
  Measuring hunger and satiety (from 0mm - 100mm)
  Choosing 0mm means less feeling of the hunger/satiety asked while choosing 100mm means more feeling of the hunger/satiety asked.

SECONDARY OUTCOMES:
Change from Baseline BMI at 3 weeks | 3 weeks
  Measuring BMI
Change from Baseline waist circumference at 3 weeks | 3 weeks
  Measuring waist circumference
Change from Baseline body composition at 3 weeks | 3 weeks
  Measuring waist circumference body composition

CONTACTS AND LOCATIONS:
Overall Officials: Seliz Bağcılar, Lecturer, Principal Investigator — Cyprus International University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akyol A, Ayaz A, Inan-Eroglu E, Cetin C, Samur G. Impact of three different plate colours on short-term satiety and energy intake: a randomized controlled trial. Nutr J. 2018 Apr 21;17(1):46. doi: 10.1186/s12937-018-0350-1. PMID 29679981
- [Result] Alblas MC, Mollen S, Fransen ML, van den Putte B. Food at first sight: Visual attention to palatable food cues on TV and subsequent unhealthy food intake in unsuccessful restrained eaters. Appetite. 2020 Apr 1;147:104574. doi: 10.1016/j.appet.2019.104574. Epub 2019 Dec 23. PMID 31877342
- [Result] Libotte E, Siegrist M, Bucher T. The influence of plate size on meal composition. Literature review and experiment. Appetite. 2014 Nov;82:91-6. doi: 10.1016/j.appet.2014.07.010. Epub 2014 Jul 15. PMID 25049139